CLINICAL TRIAL: NCT06794034
Title: Efficacy of taVNS Versus Sham Stimulation in Reduing Depressive Symptoms in Patients With Epilepsy: a Multi-center, Double-blinded, Randomized, 20-week, Parallel-arm, Superiority Study
Acronym: TIDES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other); Ningbo Medical Center Lihuili Hospital (Other Government); First Affiliated Hospital of Zhejiang University (Other); Jinhua Second Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-0182
Record Dates: First submitted 2024-11-17; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-11

CONDITIONS: Depressive Symptoms in Patients With Epilepsy
Keywords: transcutaneous auricular vagus nerve stimulation; epilepsy; depression
MeSH Terms: conditions — Epilepsy; Depression | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Intervention arm: taVNS 25Hz+routine treatment, three times daily, 30 mins Sham arm: taVNS 1Hz+routine treatment, three times daily, 30 mins
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The device provider assigns the device directly to the patient for training and use after allocation. All the scales will be assessed by the same site assessor, who has undergone consistency training. The doctors, patients, scale assessors and statisticians are all blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "xinlepai","taVNS" 25Hz (Experimental): The "xinlepai", a transcutaneous auricular vagus nerve stimulator (taVNS), was used with a stimulation frequency of 25Hz, combined with conventional treatment. Use 3 times daily for 30 minutes each time.
  Interventions: Device: Intervention
- "xinlepai","taVNS" 1Hz (Sham Comparator): The "xinlepai", a transcutaneous auricular vagus nerve stimulator (taVNS), was used with a stimulation frequency of 1Hz, combined with conventional treatment. Use 3 times daily for 30 minutes each time.
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: Intervention — taVNS 25Hz+routine treatment, three times daily, 30 mins
  Arms: "xinlepai","taVNS" 25Hz
Device: Sham Comparator — taVNS 1Hz+routine treatment, three times daily, 30 mins
  Arms: "xinlepai","taVNS" 1Hz

SUMMARY:
The purpose of this study is to compare the efficacy of taVNS versus sham stimulation in reduing depressive symptoms in patients with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Adults age ≥18
* Confirmed diagnosis of epilepsy (based on 2014 definition by ILAE)
* Having comorbidity with mild-moderate depression (confirmed diagnosis by a psychiatrist)
* Willing and able to provide informed conset

Exclusion Criteria:

* Those experiencing status epilepticus or frequent seizures requiring emergency medication within the year prior to recruitment
* Those with severe depression or anxiety who are in urgent need of psychiatric care
* Those who are imminently suicidal or unable to keep themselves safe
* Those experiencing severe cognitive difficulties with day-to-day memory, attention, and ability to learn basic information
* Those having a pacemaker, a invasive vagus nerve stimulator, or a metal implant
* The pinna is not suitable for earplugs
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Depression response proportion | at 20th week
  depression response proportion=(number of responders/total number of group patients)*100%, depression response defined as ≥50% reduction in HAMD-17 scores at 20th week

SECONDARY OUTCOMES:
Depression remission proportion | at 20th week
  depression remission proportion=(number of remission patients/total number of group patients)*100%, depression remission defined as HAMD-17 scores ≤ 7
Anxiety | at 20th week
  Changes in the 14-item Hamilton Anxiety Scale (HAMA-14) score from baseline.The total score of the HAMA-14 ranges from 0 to 56, with the higher the score, the more serious the anxiety.
Seizure frequency | at 20th week
  change from baseline in seizure frequency (times per week)
Seizure severity | at 20th week
  change from baseline in Liverpool Seizure Severity Scale (LSSS) scores.The total score of the LSSS ranges from 0 to 11 points, and the higher the score, the higher the severity of seizures
Sleep quality | at 20th week
  change from baseline in Pittsburgh Sleep Quality Index (PSQI) scores.The total score of PSQI ranges from 0 to 21, with the higher the score, the worse the sleep quality.
Suicidality | at 20th week
  change from baseline in the Mini-International Neuropsychiatric Interview (MINI) Suicide Risk Module scores.The MINI Suicide Risk Module has an overall score ranging from 0 to 33, with higher scores associated with higher suicide risk.
Quality of life | at 20th week
  change from baseline in quality of life in epilepsy inventory-31 scale, which has a total of 31 items divided into 7 aspects and 1 overall entry, the higher the score, the higher the quality of life.
Adverse events | at 4th 、8th、12th、16th、20th 、22th week
  patient-reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: yi guo, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (5):
- China (5):
  - The Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The First People's Hospital of Jiaxing, Jiaxing, Zhejiang
  - Jinhua Second Hospital, Jinhua, Zhejiang
  - Ningbo Medical Center Li Huili Hospital, Ningbo, Zhejiang
  - The Fourth Affiliated Hospital, School of Medicine, Zhejiang University, Yiwu, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided